CLINICAL TRIAL: NCT02357030
Title: Phase IIa Open Label Study to Evaluate the Safety, Tolerability, and Efficacy of KPAX 002 (Methylphenidate Hydrochloride + K-PAX Synergy) as a Treatment for Gulf War Illness in Patients Meeting the Kansas Case Definition
Brief Title: Methylphenidate Plus GWI-Nutrient Formula as a Treatment for Patients With Gulf War Illness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: K-PAX Pharmaceuticals, Inc. (Industry)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-PAX-002-2; CDMRP- GW130047 (Other: CDMRP)
Record Dates: First submitted 2015-01-25; First posted 2015-02-06 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; nutrients; methylphenidate; mitochondria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methyl-P plus GWI Nutrient Formula (Experimental): Methylphenidate hydrochloride plus a GWI Nutrient Formula (K-PAX Synergy), both taken twice daily.
  Interventions: Drug: Methyl-P plus GWI Nutrient Formula

INTERVENTIONS:
Drug: Methyl-P plus GWI Nutrient Formula — Week 1:
  * One tablet of Methyl-P (5mg) twice daily
  * Four tablets of GWI Nutrient Formula twice daily
  Week 2 to Week 12 :
  * Two tablets of Methyl-P (10mg) twice daily
  * Four tablets of GWI Nutrient Formula twice daily
  Other Names: KPAX 002

SUMMARY:
The Gulf War Synergy Trial will evaluate the safety and efficacy of a currently available medication, methylphenidate (Ritalin®), combined with a GWI Nutrient Formula (K-PAX Synergy) to treat Gulf War Illness (GWI).

DETAILED DESCRIPTION:
This trial will evaluate the safety and efficacy of a currently available medication, methylphenidate (Ritalin®), combined with a mitochondrial support nutrient formula (K-PAX Synergy) to treat Gulf War Illness (GWI).

The nutrient formula to be used in this trial is a broad-spectrum micronutrient supplement. This nutrient formula provides GWI patients with vitamins, minerals, and other cofactors (amino acids, antioxidants, and mitochondrial cofactors) to complement the low-dose Central Nervous System (CNS) stimulant (methylphenidate). The low-dose CNS stimulant provides the necessary catalyst to augment the metabolism of cellular fuel and the production of cellular energy.Therapeutic dosages of micronutrients are provided to support the functioning of the nervous, endocrine, and immune systems to a level at which a lower than customary dosage of methylphenidate can produce positive clinical effects on GWI symptoms and also be well tolerated without further depleting or degrading these systems.

The dose of methylphenidate (Ritalin®) being tested in this study is relatively low (5-10mg twice daily). This drug has been in clinical use for over 50 years for the treatment of Narcolepsy and Attention Deficit Disorder and has a well-described safety profile when used as recommended. GWI and Chronic Fatigue Syndrome (CFS) share a high degree of symptom overlap. They have both been linked to mitochondrial dysfunction. Methylphenidate alone has been studied as a treatment for CFS in the past and has been shown to produce mild benefits and be well-tolerated. When provided as innovative therapy, methylphenidate plus this CFS Nutrient Formula has produced substantial improvements in CFS symptoms in a limited number of patients, and demonstrated excellent tolerability.

Use of low dose methylphenidate coadministered with a mitochondria support nutrient formula has not been previously evaluated in a controlled clinical study. The risk to patients using this combination is believed to be low, especially in the context of a well-controlled clinical study. Furthermore, this combination is not expected to increase the incidence or severity of adverse events associated with methylphenidate.

ELIGIBILITY:
1. Male and female patients between the ages of 18 and 64, inclusive at the time of informed consent
2. Patients who currently meet the Kansas Case Definition for GWI
3. Patients who are otherwise in good health based on medical history and screening evaluation as determined by Investigator (see below for specific exclusion criteria)
4. Willingness to not take any multivitamin, nutritional or herbal supplements other than the study treatment during the course of the trial; at least a one week washout of current nutritional supplements will be required between the screening and baseline visits. Nutritional supplements that are exempted from this requirement are limited to the following (other exemptions require a waiver by the Medical Monitor):

   1. Probiotic supplements (L. acidophilus, Bifidobacterium, etc.)
   2. Fiber supplements
   3. Fish oil supplements
   4. Digestive enzymes
   5. Melatonin < 10mg per day
   6. Calcium < 600mg per day
   7. Magnesium < 400mg per day
   8. Vitamin D < 400 i.u. per day
5. Willingness to not consume any caffeine-containing supplements during the study period (coffee, tea and chocolate are exempt). These supplements include but are not limited to the following:

   1. Red Bull®
   2. Monster®
   3. Rockstar®
   4. 5-hour® energy shots
6. Willingness to not consume any prescription stimulants (i.e. Provigil®, Nuvigil®, Adderall®, Ritalin®, amphetamines) during the study period.
7. Willingness to not consume any pseudoephedrine-containing products during the study period.
8. Willingness of females to practice effective contraception.

Exclusion Criteria:

1. Pregnancy or lactation
2. Active substance or alcohol abuse and/or a history of prescription stimulant abuse
3. Hospitalization within the past five years for any of the following:

   1. Active substance or alcohol abuse and/or a history of prescription stimulant abuse
   2. Major Depressive Disorder (MDD)
   3. Post Traumatic Stress Disorder (PTSD)
4. Previous or current diagnosis of schizophrenia or bipolar disorder
5. Currently taking any prescription medication to treat anxiety on a daily basis
6. Use of any of the below medications more than 3 times per week within the past 3 months:

   1. MAO inhibitors
   2. Anti-psychotic medications
   3. Prescription stimulants (i.e. Provigil®, Nuvigil®, Adderall®, Ritalin®, or any other amphetamines)
   4. Coumarin anticoagulants (Coumadin®)
7. Daily concurrent use of more than one antidepressant medication except if one of the two antidepressant medications are one of the following (unless specifically granted a waiver by the Medical Monitor):

   1. Amitriptyline ≤ 100 qhs
   2. Trazodone ≤ 100 qhs
   3. Doxepin ≤ 50 qhs
8. Active medical conditions including:

   1. Glaucoma
   2. Diabetes mellitus
   3. Current stomach or duodenal ulcer
   4. Uncontrolled hypertension (blood pressure at screening of systolic >160 or diastolic >90)
   5. Heart disease (including a history of cardiac arrhythmia, cardiac ischemia, syndrome of Torsade de Pointes, myocardial infarction or cerebrovascular event)
   6. Motor tics or a diagnosis or family history of Tourette's syndrome
   7. Previous history of seizures
   8. A diagnosis of any of the following conditions:

      * Cancer (receiving systemic treatment either currently or within the past 12 months)
      * Chronic Renal Disease
      * Chronic Liver Disease
      * HIV Infection
      * Chronic Hepatitis B or C
      * Systemic Lupus Erythematosus
      * Multiple Sclerosis
      * Rheumatoid Arthritis
      * Parkinson's Disease
      * Amyotrophic Lateral Sclerosis (ALS)
      * Any chronic infectious disease lasting six months or longer
9. Clinically significant laboratory test values as determined by the Medical Monitor
10. Clinically significant ECG abnormalities as determined by the Medical Monitor
11. The taking of another investigational treatment either currently or within 30 days of the screening visit
12. Compliance criteria: A subject will not be eligible if he/she, in the opinion of the Investigator, will be unable to comply with any aspect of this study protocol, including the visit schedule.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported Checklist Individual Strength (CIS) total score | Week 12

SECONDARY OUTCOMES:
Percentage of patients with 20% or greater improvement in the CIS total score | Week 12
Concentration Disturbances Subscore on the CIS | Week 12
Concentration Disturbances Score by Visual Analog Scale (VAS) | Week 12
Fatigue Score by Visual Analog Scale (VAS) | Week 12
Pain Score by Visual Analog Scale (VAS) | Week 12
Sleep Score by Visual Analog Scale (VAS) | Week 12
Mitochondrial Function Assays | Week 12
GWI Symptoms Assessment Tool (SAT) Score | Week 12
Number of Participants with Adverse Events to Assess Safety and Tolerability | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jon D. Kaiser, MD, Study Director — K-PAX Pharmaceuticals, Inc.; Mark Holodniy, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- Veterans Administration Palo Alto Health Care System (VAPAHCS), Palo Alto, California, United States